CLINICAL TRIAL: NCT06512155
Title: The Effect of Pregabalin on Perioperative Sleep Quality in Orthopedic Surgery Patients: a Prospective, Randomized, Controlled Study
Brief Title: Improving Perioperative Sleep Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mengchang Yang (Other)
Responsible Party: Sponsor-Investigator, Mengchang Yang, Doctor, Sichuan Provincial People's Hospital
Organization: Sichuan Provincial People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sleep disorders-1
Record Dates: First submitted 2024-06-24; First posted 2024-07-22 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-07

CONDITIONS: Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Pregabalin; Zolpidem

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pregabalin Group (Experimental): The Pregabalin group started taking Pregabalin 75mg bid two days before surgery and Pregabalin 150mg bid from the day before surgery to three days after surgery
  Interventions: Drug: Pregabalin
- Zolpidem Group (Experimental): Patients in the zolpidem group took zolpidem 10mg every night from two days before surgery to three days after surgery
  Interventions: Drug: Zolpidem
- Control group (No Intervention): Control group patients do not take any additional medication that affects sleep

INTERVENTIONS:
Drug: Pregabalin — Start taking 75mg bid of pregabalin two days before surgery, and take 150mg bid of pregabalin from one day before surgery to three days after surgery
  Other Names: Pregabalin Capsules (Lerika)
  Arms: Pregabalin Group
Drug: Zolpidem — Take zolpidem 10mg qn from two days before surgery to three days after surgery
  Other Names: Zolpidem Tartrate Tablets（Sinuosi）
  Arms: Zolpidem Group

SUMMARY:
In today's day of increasing surgical volume, perioperative sleep disorders are an issue that cannot be ignored. They are an important component of perioperative brain protection. Physiologically and psychologically, sleep disorders cause serious damage to patients. The application of pregabalin aims to improve the sleep quality of hand surgery patients, and its anti anxiety effect can also alleviate preoperative anxiety. At the same time, its analgesic mechanism is different from that of opioid drugs, which is also conducive to reducing the use of opioid drugs. Therefore, we propose the following hypothesis: for orthopedic patients with high incidence of postoperative pain and sleep disorders, the use of pregabalin will improve the perioperative sleep quality of such patients.To test the above hypothesis, our research group plans to conduct this prospective, randomized, positive control study.

DETAILED DESCRIPTION:
Perioperative sleep disorders mainly refer to the syndrome in which patients undergoing surgery experience disrupted sleep wake rhythms before and/or after surgery, leading to abnormal sleep quality or behavior during sleep. Clinical manifestations include fragmented sleep, easy awakening at night, difficulty falling asleep, insufficient sleep time, early bedtime, or disrupted sleep rhythm at least one day before or after surgery. The latest meta-analysis study indicates that the incidence of preoperative sleep disorders in surgical patients is as high as 60%. After surgery, about 60-70% of patients will have postoperative sleep disorder (PSD), and even 23% of patients will have sleep disorder until the fourth day after surgery. Among various surgeries, orthopedic surgery has a high incidence of PSD due to its long operation time and wide surgical range. In the study by Duan G and colleagues, the PSD incidence rate of spinal orthopedic surgery in orthopedics was 35.4%, and the PSD incidence rate of limb surgery was 27%.

Sleep disorders may lead to a range of complications, including cognitive impairment, delayed postoperative recovery, acute pain, and cardiovascular accidents. In the hospital environment, factors that lead to poor sleep include pain, anxiety, noise, interference from hospital staff, continuous ambient lighting, and uncomfortable beds; After completing the surgery, factors such as the size of the surgery, the use of opioid drugs, inflammatory mediators, the release of various hormones, and pain contribute to a high incidence of sleep disorders, with pain being the most common cause, and there is an interactive relationship between postoperative sleep disorders and pain. It is worth noting that patients with poor preoperative sleep quality have a higher probability of developing sleep disorders after surgery. Therefore, it is necessary to comprehensively consider these factors and take corresponding preventive measures to reduce the incidence of perioperative sleep disorders.

According to the sleep care guidelines, for postoperative patients entering the ICU, maintaining a quiet and dim environment and reducing interruptions in nighttime care activities are recommended to improve sleep quality and efficiency. A meta-analysis shows that the use of earplugs and eye masks also helps promote sleep in ICU patients. However, it is evident that this method is not suitable for patients who are admitted to regular multi person wards after surgery. Although in a meta-analysis, there was insufficient evidence to suggest that drug therapy can improve the quality or quantity of sleep in patients with poor postoperative sleep. Even compared to placebo or no treatment, there is no established drug category or specific drug that is superior to placebo or no treatment [6]. However, drug therapy is still widely used for patients with perioperative sleep disorders due to its convenience, strong feasibility, and high patient acceptance.

In current clinical practice, the main drugs used to address perioperative sleep disorders are sleeping pills and painkillers. Specifically, sleeping pills are mainly divided into first generation, second generation, and third generation sedative hypnotic drugs. These drugs mainly exert extensive inhibition on the central nervous system, causing it to transition from an excited state to an inhibited state. However, their effect on improving sleep structure is not satisfactory, especially the second-generation drugs - benzodiazepines, which can change the usual sleep pattern, prolong shallow sleep, shorten the duration of REM sleep, and delay the appearance of the first REM sleep. This change, which is similar to the postoperative sleep structure, is more detrimental to the improvement of patients' sleep, therefore the effect is not satisfactory. As for painkillers, opioids are the most commonly used class in clinical practice. Even though they have strong analgesic effects, they have been found to dose dependently inhibit REM and SWS sleep in normal volunteers and animal experiments. In addition, in Cronin AJ et al.'s study, postoperative patients suffered from severe sleep disorders even when avoiding opioid use and pain was well controlled. Therefore, the improvement of sleep in perioperative patients cannot be limited to the use of the above two drugs.

Pregabalin is a gabapentin class drug that inhibits the influx of calcium ions into the presynaptic membrane of neurons and reduces the release of excitatory neurotransmitters (including glutamate, aspartic acid, substance P, calcitonin gene-related peptide, norepinephrine, serotonin, dopamine, etc.) by binding to the α 2 δ pressure group containing voltage-gated calcium channels. Its analgesic, anti anxiety, and anticonvulsant effects are widely used in various clinical diseases. Pregabalin has been approved for the treatment of neuropathic pain and partial seizures in the United States and Europe. It can also be used for fibromyalgia in the United States and for the treatment of generalized anxiety disorder in Europe. While treating patients with this type of chronic disease, its effect on improving sleep has been discovered. Studies have found that pregabalin exhibits significant sleep improvement effects from the initial stage of medication, and its therapeutic efficacy is maintained throughout the entire treatment phase. Similar sleep improvement effects to alprazolam have also been found in normal healthy individuals. The mechanism by which pregabalin improves sleep is still unclear, and it is speculated to be related to its ability to reduce excitatory neurotransmitters. Currently, there is no relevant research on the impact of pregabalin on sleep quality in perioperative patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤ Age ≤ 65 years old, gender unlimited.
* ASA level I-II.
* Plan to undergo elective total knee arthroplasty, total hip arthroplasty, and spinal vertebral body surgery.

Exclusion Criteria:

* Patients with preoperative sleep problems.
* Patients refuse to participate in the study.
* The patient has any allergies or contraindications to the drugs used in the study.
* The patient has a history of long-term use of medications such as pregabalin or gabapentin.
* The patient has a history of long-term use of any painkillers or sleeping pills.
* The patient has cognitive impairment and is unable to conduct visits and communication.
* The patient has a history of renal dysfunction or any other serious organ dysfunction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-26 (Actual)

PRIMARY OUTCOMES:
Athens Insomnia Scale | From the second day of medication to five days after surgery
  The Athens Insomnia Scale has a minimum score of zero and a maximum score of 24. When the score is greater than or equal to 6, it indicates the presence of sleep disorders, and the higher the score, the more severe the sleep disorders.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index score | On the 30th day after surgery
  The total score range of the Pittsburgh Sleep Quality Index is 0-21 points. The higher the score, the worse the sleep quality. An index greater than or equal to 8 points is considered to have a sleep quality issue
Hamilton Anxiety Scale (HAMA) | Two days before surgery and five days after surgery
  A total score of ≥ 29 on the Hamilton Anxiety Scale may indicate severe anxiety 21 points, there must be obvious anxiety; ≥ 14 points, there must be anxiety; Exceeding 7 points may indicate anxiety; If it is less than 7 points, there are no symptoms of anxiety.
VAS score | Five days after surgery
  Evaluate patient pain using VAS score five days after surgery
Perioperative opioid consumption | Immediately after discharge
  Perioperative opioid consumption, converted to morphine equivalent
Postoperative hospitalization time | Immediately after discharge
  Postoperative hospitalization time
The incidence of various adverse events | Immediately after discharge
  The incidence of various adverse events, including fatigue, drowsiness, dizziness, nausea and vomiting, blurred vision, and other psychological symptoms such as hallucinations, agitation, nightmares, depression, etc
Patient satisfaction survey | Immediately after discharge
  The patient satisfaction survey during hospitalization is divided into four levels: very satisfied, relatively satisfied, relatively dissatisfied, and very dissatisfied.
Hamilton Depression Scale（HAMD） | Two days before surgery and five days after surgery
  Hamilton Depression Scale total score<7: normal; A total score of 7-17 indicates possible depression; A total score of 17-24 points indicates the presence of depression; Total score>24: Severe depression。

CONTACTS AND LOCATIONS:
Overall Officials: Yang Mengchang, Doctor, Principal Investigator — Sichuan Provincial People's Hospital
Locations (1):
- Sichuan Provincial People's Hospita, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No